CLINICAL TRIAL: NCT06945302
Title: The Effect of Inulin Supplementation on Nutritional Status, Anthropometric Measurements and Bowel Symptoms in Individuals With IBS-C: RCT
Brief Title: The Effect of Inulin Supplementation in Individuals With IBS-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mardin Artuklu University (Other)
Responsible Party: Principal Investigator, Çağlar Akçalı, Assist. Prof., Mardin Artuklu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-377
Record Dates: First submitted 2025-04-07; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Inulin; IBS (Irritable Bowel Syndrome); Nutritional Status; Anthropometric Measurement
Keywords: Anthropometric measurements; bowel symptoms; inulin; irritable bowel syndrome; nutritional status
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Individuals were randomly assigned to one of two groups: Intervention (n=17) and control (n=17) groups.
Who Masked: Participant
Masking Description: Participants were blinded to groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): products containing a total of 9.2 g (4.6 g twice a day) inulin/oligofructose (50/50) mixture (prebiotic group) that individuals should consume daily were delivered to individuals in identical opaque bags.
  Interventions: Dietary Supplement: Intervention Group
- Control (Placebo Comparator): products containing a total of 9.2 g (4.6 g twice a day) maltodextrin (placebo group) that individuals should consume daily were delivered to individuals in identical opaque bags
  Interventions: Dietary Supplement: Control group (placebo)

INTERVENTIONS:
Dietary Supplement: Intervention Group — products containing a total of 9.2 g (4.6 g twice a day) inulin/oligofructose (50/50) mixture (prebiotic group) that individuals should consume daily were delivered to individuals in identical opaque bags.
  Arms: Intervention group
Dietary Supplement: Control group (placebo) — products containing a total of 9.2 g (4.6 g twice a day) maltodextrin (placebo group) that individuals should consume daily were delivered to individuals in identical opaque bags.
  Arms: Control

SUMMARY:
Background: This study aimed to evaluate the effects of inulin supplementation on nutritional intake, anthropometric parameters, and bowel symptoms in individuals diagnosed with IBS-C.

Method: This was a randomised, single-blind, placebo-controlled clinical trial. Participants were randomly allocated into intervention (inulin) and control (placebo) groups for 8 weeks. Assessments included dietary intake, anthropometric measurements, and IBS symptoms.

DETAILED DESCRIPTION:
Irritable Bowel Syndrome (IBS) is a common functional gastrointestinal disorder characterised by chronic abdominal pain, bloating, and altered bowel habits, often without identifiable organic pathology. IBS with predominant constipation (IBS-C) presents management challenges due to its multifactorial aetiology and impact on quality of life.

Inulin, a naturally occurring prebiotic dietary fibre found in many plants, has been studied for its beneficial effects on gut health, bowel function, and body composition. It may increase short-chain fatty acid production, improve intestinal transit, and promote beneficial gut microbiota such as Bifidobacteria. However, evidence on the specific benefits of inulin supplementation in individuals with IBS-C remains limited.

Inclusion criteria were being between the ages of 19-65 years, volunteering to participate in the study, being diagnosed with IBS by a physician according to Rome IV criteria, and having two of the three criteria according to Rome IV criteria: associated with defecation (alleviation), associated with change in defecation frequency, associated with change in stool appearance / symptoms started at least 6 months before the diagnosis was made and recurrent abdominal pain at least 1 day a week for the last 3 months. Exclusion criteria were a history of gastrointestinal surgery (except appendectomy and cholecystectomy), inflammatory bowel disease, lactose malabsorption, gastroenteritis, celiac disease, gastric and duodenal ulcer, metabolic diseases (cardiac, hepatic and renal diseases, diabetes, etc.), malignancy. ), history of malignancy, pregnancy and lactation, use of intestinal motility and antidepressant drugs, involuntary body weight loss of more than 5 kg in the last 3 months, use of dietary fibre supplements in the last 3 months, use of antibiotics in the last 3 months, and use of prebiotic and probiotic supplements in the last 3 months.

In this study, eligible participants were randomly allocated into two groups:

* Intervention group (n=17): received 9.2 g/day of an inulin-oligofructose mixture (50:50), split into two doses daily.
* Control group (n=17): received an isocaloric placebo (maltodextrin, 9.2 g/day) using the same dosing schedule.

The intervention period was 8 weeks, during which participants continued their usual dietary habits. Assessments included dietary intake evaluations, anthropometric measurements (weight, BMI, waist and hip circumference, body composition via bioelectrical impedance), and IBS symptoms (using the IBS-SSS) at baseline and after 8 weeks.

The primary outcome was the change in IBS symptom severity (IBS-SSS scores). Secondary outcomes were changes in anthropometric parameters and dietary intake.

ELIGIBILITY:
Inclusion Criteria:

* the individuals were between 19-65 years of age
* volunteer to participate in the study
* Individuals diagnosed with IBS by a physician according to Rome IV criteria

Exclusion Criteria:

* a history of gastrointestinal surgery (except appendectomy and cholecystectomy)
* inflammatory bowel disease
* lactose malabsorption
* gastroenteritis
* celiac disease
* gastric
* duodenal ulcer
* metabolic diseases (cardiac, hepatic and renal diseases, diabetes, etc.)
* history of malignancy
* pregnancy and lactation
* use of intestinal motility
* antidepressant drugs
* involuntary body weight loss of more than 5 kg in the last 3 months
* use of dietary fibre supplements in the last 3 months
* use of antibiotics in the last 3 months
* use of prebiotic and probiotic supplements in the last 3 months.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2022-01-03 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Irritable Bowel Syndrome - Symptom Severity Score/(IBS-SSS) | 8 week
  The IBS-SSS scale was used to assess the severity of irritable bowel syndrome symptoms. This scale consists of a total of 5 questions, each of which is scored between 0 and 100. The questions provide information about the severity and frequency of abdominal pain, the severity of abdominal distension, the level of satisfaction with bowel habits and the impact of the disease on quality of life. An increase in the score obtained from the scale indicates an increase in symptom severity. ROC (Receiver Operating Characteristic) analysis was applied for the cut-off point of the scale. Accordingly, the cut-off point was calculated as 217.5.

SECONDARY OUTCOMES:
Outcome Measure 1: Height Measurement | 8 weeks
  Description: "The height of the participants was measured using an inflexible tape measure with their head, hips, and heels touching the wall, and their feet standing side by side and in the Frankfort plane."
  * Unit: centimeters
Outcome Measure 2: Waist Circumference | 8 weeks
  Description: "The waist circumference was measured using a non-flexible tape measure with a sensitivity of 0.1 cm at the midpoint between the iliac crest and the lowest rib margin."
  * Unit: centimeters
Outcome Measure 3: Hip Circumference | 8 weeks
  Description: "Hip circumference was measured at the widest point of the hips using a non-flexible tape measure."
  * Unit: centimeters
Outcome Measure 4: Lean Body Mass | 8 weeks
  Description: "Lean body mass (kg) assessed using bioelectrical impedance analysis (Tanita BC 601)."
  * Unit: kilograms
Outcome Measure 5: Body Fat Percentage | 8 weeks
  Description: "Body fat percentage (%) assessed via bioelectrical impedance analysis (Tanita BC 601)."
  * Unit: percentage (%)
Outcome Measure 6: Total Body Water | 8 weeks
  Description: "Total body water percentage (%) assessed via bioelectrical impedance analysis (Tanita BC 601)."
  * Unit: percentage (%)
Outcome Measure 7: Bone Mass | 8 weeks
  Description: "Bone mass (kg) assessed using bioelectrical impedance analysis (Tanita BC 601)."
  * Unit: kilograms
Outcome Measure 8: BMI | 8 weeks
  Description: "Body mass index calculated from height and weight measurements (kg/m²)."
  * Unit: kg/m²
Determination of Nutrient Consumption Status | 8 week
  In order to determine the nutritional status of the participants, 24-hour food consumption records were taken at the beginning of the study and one-day food consumption records were taken in the 8th week. In determining the ingredients and quantities of some of the meals consumed, the book 'Standard Recipes' was used. The meals cooked at home were calculated by asking questions. 'Food and Nutrient Photo Catalogue' was used in order to evaluate the consumption measurements and quantities of foods accurately. The calculation of energy, macro and micronutrient values of the foods consumed was done with the Computer Assisted Nutrition (BEBIS) programme.

CONTACTS AND LOCATIONS:
Locations (1):
- Mardin Artuklu University, Mardin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy concerns and ethical considerations related to the small sample size, which may increase the risk of participant identification

REFERENCES:
- [Result] Merdol, T.K. (2011). Standard meal schedules for institutions (4. edt). Ankara: Hatipoğlu Publishing.
- [Result] Rakıcıoğlu, N., Acar Tek, N., Ayaz, A., Pekcan, G. (2012). Food and nutrient photo catalog. Ankara: Hatiboğlu Publishing.
- [Result] World Health Organization (WHO). (2011). Waist circumference and waist-hip ratio: report of a WHO expert consultation, Geneva, 8-11 December 2008.
- [Result] Bjelica, D., Popović, S., Kezunović, M., Petković, J., Jurak, G., & Grasgruber, P. (2012). Body height and its estimation utilising arm span measurements in Montenegrin adults. Anthropological Notebooks, 18(2).